CLINICAL TRIAL: NCT03045172
Title: A Double Blind Placebo Controlled Trial of Autologous Platelet Rich Plasma (PRP) Intradermal Injections for the Treatment of Vulvar Lichen Sclerosus
Brief Title: Platelet Rich Plasma (PRP) for Vulvar Lichen Sclerosus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Center for Vulvovaginal Disorders (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GCRF-1
Record Dates: First submitted 2017-02-01; First posted 2017-02-07 (Estimated); Last update posted 2018-10-25 (Actual); Status verified 2018-10

CONDITIONS: Lichen Sclerosus of Vulva
Keywords: Lichen Sclerosus; Platelet Rich Plasma; Vulvar; Vulva
MeSH Terms: conditions — Vulvar Lichen Sclerosus; Lichen Sclerosus et Atrophicus

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Dermatopathologist
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): 20 subjects with Platelet Rich Plasma injections
  Interventions: Biological: Platelet Rich Plasma
- Group 2 (Placebo Comparator): 10 subjects with placebo injections
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Platelet Rich Plasma — PRP
  Arms: Group 1
Drug: Placebo — Saline
  Arms: Group 2

SUMMARY:
Lichen sclerosus (LS) is a skin condition of the external genitals (vulva) of women. LS causes vulvar itching, pain, and burning. In addition, LS causes scarring of the vulva which may cause significant sexual dysfunction or pain. Lastly, 4-6% of women with LS will develop vulvar cancer.

The current "gold standard" treatment for lichen sclerosus is potent steroids creams. When used correctly, steroid creams help to decrease the symptoms of itching and burning and can prevent further vulvar scarring. In addition, proper treatment reverses the underlying inflammation of LS, and may lower the risk of getting cancer. While useful, steroid creams may have serious side effects that include thinning of the skin, fungal infections, and lowering the immune system.

Platelet-rich plasma (PRP) is a platelet concentrate that helps to speed up tissue healing, without serious side effects, in a very wide range of medical conditions such as diabetic foot ulcers, muscle injury, tendon injury, and in a variety of cosmetic procedures. The PRP works because of its high level of proteins that help with wound healing. It is also apparent from the majority of published studies that PRP therapy has minimal risk of scar tissue formation or significant bad side effects.

Recently, there was an exploratory study of twelve subjects that used PRP for the study treatment of lichen sclerosus. While this study showed good success, the study was limited because of its small size and lack of placebo (a drug or study treatment that contains no active ingredient) control.

DETAILED DESCRIPTION:
This will be a randomized single-blind placebo controlled trial to evaluate the efficacy and safety of autologous Platelet-rich Plasma (PRP) for the treatment of vulvar lichen sclerosus. Thirty patients with a diagnosis of biopsy proven active vulvar lichen sclerosus will be recruited from one center. This study will consist of a two-week screening period and a 12-week treatment period. At the beginning of the screening period, a 4 millimeter punch skin biopsy sample will be collected from each patient to confirm the diagnosis of active lichen sclerosus and to rule out the diagnoses of lichen planus, psoriasis, candidiasis, and vulvar intraepithelial neoplasia. In addition, vulvoscopy will be performed at the screening visit and after the 12-week treatment period to rule out vulvar carcinoma. All eligible patients will be randomized to receive either placebo (saline injections) (10 subjects) or two separate treatments of PRP separated by 6 weeks (20 subjects). Each treatment would consist of an injection of 5 ml of autologous platelet-rich plasma (PRP) injected subdermally and intra-dermally, infiltrating the areas of the vulva affected by active lichen sclerosus. A repeat biopsy will be performed adjacent to the original biopsy site at the 12 week visit.

The preparation of autologous PRP is as follows: 60 cc of whole blood will be removed via venopuncture. Preparation of PRP is done using a proprietary, FDA approved, centrifuge which uses a laser and a closed sterile system to identify and isolate the most platelet rich fraction of 60ml of whole blood. [Magellan® Autologous Platelet Separator System. Arteriocyte Medical Systems. Hopkinton, MA USA].

The PRP will be collected in a blackened syringe so that neither Dr. Goldstein (the physician administering the PRP) nor the patient will know if she is receiving the PRP or placebo.

After isolation of the PRP, calcium chloride (0.7ml) will be added to the 5 ml of PRP isolate to activate the thrombin cascade, thereby causing degranulation of platelets, releasing growth factors and cytokines, and starting the transformation of the PRP to platelet rich fibrin matrix (PRFM).

The primary efficacy variable will be performed by a blinded dermatopathologist who will evaluate the inflammatory infiltration on biopsy specimens obtained during the screening period and at the Week 14 visit (1 to 4 scales). A secondary endpoint will be changes from baseline in the "Clinical Scoring System for Vulvar Lichen Sclerosus" (CSS) a validated instrument that assessment both an investigator's impression of the severity of disease and a patient's impression of the severity of her disease.

All adverse events will be recorded, including serious adverse events. A physical examination will be performed at each visit.

ELIGIBILITY:
Inclusion Criteria:

* Female, 18 year or older
* With a diagnosis of biopsy proven active vulvar lichen sclerosus
* Signed written informed consent
* Willingness and ability to comply with the study requirements
* Subject must have a score of 5 or greater in the itching (pruritus) domain of the CSS upon enrollment

Exclusion Criteria:

* Who have received systemic immunosuppressants (e.g. corticosteroids) within 12 weeks prior to participation in the study
* Who have been treated with topical therapy (e.g. topical corticosteroids, topical calcineurin inhibitors, topical estrogen, topical testosterone) at the affected area within 16 weeks prior to participation in the study.
* Who are immunocompromised (e.g. lymphoma, AIDS, Wiskott-Aldrich Syndrome) or have an uncontrolled malignant disease
* Who suffer from systemic of generalized infections (bacterial, viral, or fungal)
* Who have been diagnosed with lichen planus, psoriasis, candidiasis, intraepithelial neoplasia, or carcinoma of the vulva
* Who had received an investigational drug within four weeks prior to the study or who intend to use other investigational drugs during the course of this study.
* Patients with severe medical conditions(s) that in the view of the investigator prohibits participation in the study.
* Who have a history of substance abuse of any factor, which limits the subject's ability to cooperate in the study procedure
* Who are uncooperative, known to miss appointments (according to subjects' records) and are unlikely to follow medical instructions pr are not willing to attend regularly scheduled visits.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 29 (Actual)
Dates: Start 2016-11; Primary Completion 2018-08 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Clinical Scoring System for Vulvar Lichen Sclerosus | 14 weeks
  A validated instrument that assesses both the investigator's impression of the severity of disease and a patient's impression of the severity of her disease pre and post-intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew T Goldstein, MD, Principal Investigator — The Center for Vulvovaginal Disorders
Locations (1):
- The Center for Vulvovaginal Disorders, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pierard GE, Pierard-Franchimont C, Ben Mosbah T, Arrese Estrada J. Adverse effects of topical corticosteroids. Acta Derm Venereol Suppl (Stockh). 1989;151:26-30; discussion 47-52. PMID 2624063
- [Background] Lubach D, Rath J, Kietzmann M. Steroid-induced dermal thinning: discontinuous application of clobetasol-17-propionate ointment. Dermatology. 1992;185(1):44-8. doi: 10.1159/000247402. PMID 1638070
- [Background] Cherian MP, AbdulJabbar M. Cushing's syndrome and adrenal suppression from percutaneous absorption of clobetasol propionate in infants. Saudi Med J. 2001 Dec;22(12):1139-41. No abstract available. PMID 11802195
- [Background] Furue M, Terao H, Rikihisa W, Urabe K, Kinukawa N, Nose Y, Koga T. Clinical dose and adverse effects of topical steroids in daily management of atopic dermatitis. Br J Dermatol. 2003 Jan;148(1):128-33. doi: 10.1046/j.1365-2133.2003.04934.x. PMID 12534606
- [Background] Sarvajnamurthy S, Suryanarayan S, Budamakuntala L, Suresh DH. Autologous platelet rich plasma in chronic venous ulcers: study of 17 cases. J Cutan Aesthet Surg. 2013 Apr;6(2):97-9. doi: 10.4103/0974-2077.112671. PMID 24023432
- [Background] Sclafani AP. Safety, efficacy, and utility of platelet-rich fibrin matrix in facial plastic surgery. Arch Facial Plast Surg. 2011 Jul-Aug;13(4):247-51. doi: 10.1001/archfacial.2011.3. Epub 2011 Feb 21. PMID 21339469
- [Background] Chen L, Yang X, Huang G, Song D, Ye XS, Xu H, Li W. Platelet-rich plasma promotes healing of osteoporotic fractures. Orthopedics. 2013 Jun;36(6):e687-94. doi: 10.3928/01477447-20130523-10. PMID 23746028
- [Background] Goldstein AT, King M, Runels C, Gloth M, Pfau R. Intradermal injection of autologous platelet-rich plasma for the treatment of vulvar lichen sclerosus. J Am Acad Dermatol. 2017 Jan;76(1):158-160. doi: 10.1016/j.jaad.2016.07.037. No abstract available. PMID 27986140
- [Background] Lubkowska A, Dolegowska B, Banfi G. Growth factor content in PRP and their applicability in medicine. J Biol Regul Homeost Agents. 2012 Apr-Jun;26(2 Suppl 1):3S-22S. PMID 23648195
- [Background] Salazar-Alvarez AE, Riera-del-Moral LF, Garcia-Arranz M, Alvarez-Garcia J, Concepcion-Rodriguez NA, Riera-de-Cubas L. Use of platelet-rich plasma in the healing of chronic ulcers of the lower extremity. Actas Dermosifiliogr. 2014 Jul-Aug;105(6):597-604. doi: 10.1016/j.ad.2013.12.011. Epub 2014 Mar 12. English, Spanish. PMID 24630241
- [Background] Moraes VY, Lenza M, Tamaoki MJ, Faloppa F, Belloti JC. Platelet-rich therapies for musculoskeletal soft tissue injuries. Cochrane Database Syst Rev. 2013 Dec 23;(12):CD010071. doi: 10.1002/14651858.CD010071.pub2. PMID 24363098
- [Background] Casabona F, Priano V, Vallerino V, Cogliandro A, Lavagnino G. New surgical approach to lichen sclerosus of the vulva: the role of adipose-derived mesenchymal cells and platelet-rich plasma in tissue regeneration. Plast Reconstr Surg. 2010 Oct;126(4):210e-211e. doi: 10.1097/PRS.0b013e3181ea9386. No abstract available. PMID 20885230
- [Background] Gunthert AR, Duclos K, Jahns BG, Krause E, Amann E, Limacher A, Mueller MD, Juni P. Clinical scoring system for vulvar lichen sclerosus. J Sex Med. 2012 Sep;9(9):2342-50. doi: 10.1111/j.1743-6109.2012.02814.x. Epub 2012 Jul 3. PMID 22759453
- Available data/document: Informed Consent Form — http://www.cvvd.org/research — Click the link titled "NEW STUDY FOR LICHEN SCLEROSUS- PLATELET RICH PLASMA (PRP)- Open to new participants" to open the informed consent.